CLINICAL TRIAL: NCT02623634
Title: Effects of Different Postures and Ventilator Flow Waveforms on the Cuff Leak Test: A Prospective Cohort Study
Brief Title: Effects of Different Postures and Ventilator Flow Waveforms on the Cuff Leak Test
Status: Completed | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Huiwen Chu, Master, Beijing Chao Yang Hospital
Other Study IDs: Bei Jing Chao Yang Hospital
Record Dates: First submitted 2015-11-13; First posted 2015-12-08 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Cuff Leak Volume
Keywords: Cuff leak test, relative factors
MeSH Terms: interventions — Patient Positioning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- observation: this study measure the cuff leak volume and cuff leak ratio according to the cuff leak test with different positions and waveform,, at the same time observe the patient general condition, vital signs, oxygen saturation, cuff leak test results under different conditions and the breathing machine parameters, the diameter of the airway, the use of sedatives and hormones, after extubation stridor and intubation is happening again, the use of NPPV after extubation, patient outcomes
  Interventions: Behavioral: Position, waveform

INTERVENTIONS:
Behavioral: Position, waveform — different positions and waveform

SUMMARY:
the purpose of this study is to analyzes the factors influencing the results of cuff leak test, in order to improve the cuff leak test on the accuracy of the prediction on airway edema after extubation.

ELIGIBILITY:
Inclusion Criteria:

* Intubation less than 24 hours before amitting respiratory intensive care unit;

Exclusion Criteria:

* unstable hemodynamics;PEEP≥10cmH2O or FiO2≥0.8

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients in RICU of Beijing chaoyang hospital with tracheal intubation
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2015-10-04 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
post-extubation stridor | 48 hours
  Inspiratory stridor within 48 hours of extubation and was usually associated with respiratory distress

SECONDARY OUTCOMES:
Extubation failure due to PES | 48 hours
  the need for reintubation in the 48 hours following extubation in a patient with post-extubation stridor.

CONTACTS AND LOCATIONS:
Overall Officials: Huiwen Chu, bachelor, Study Director — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chao Yang Hospital RICU, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Prinianakis G, Alexopoulou C, Mamidakis E, Kondili E, Georgopoulos D. Determinants of the cuff-leak test: a physiological study. Crit Care. 2005 Feb;9(1):R24-31. doi: 10.1186/cc3012. Epub 2004 Nov 29. PMID 15693963
- [Result] Kemper KJ, Benson MS, Bishop MJ. Predictors of postextubation stridor in pediatric trauma patients. Crit Care Med. 1991 Mar;19(3):352-5. doi: 10.1097/00003246-199103000-00012. PMID 1999096
- [Result] Potgieter PD, Hammond JM. "Cuff" test for safe extubation following laryngeal edema. Crit Care Med. 1988 Aug;16(8):818. doi: 10.1097/00003246-198808000-00020. No abstract available. PMID 3396380
- [Result] El-Orbany M, Salem MR. Endotracheal tube cuff leaks: causes, consequences, and management. Anesth Analg. 2013 Aug;117(2):428-34. doi: 10.1213/ANE.0b013e318292ee21. Epub 2013 Jun 6. PMID 23744958